CLINICAL TRIAL: NCT06367426
Title: A Dose-blocked-randomized, Double-blind, Placebo-controlled, Single and Multiple Dosing, Dose-escalation Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics of DDN-A-0101 in Healthy Adults and Elderly Subjects
Brief Title: A Phase I Study of DDN-A-0101 in Healthy Volunteers and Elder People
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacobio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pharmacobio
Record Dates: First submitted 2024-04-02; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: To maintain double-blindness, DDN-A-0101 tablets and placebo with the same formulation and properties that cannot be distinguished in appearance will be used, and sub-packaging will also be the same.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: DDN-A-0101 for PART 1 (Experimental): DDN-A-0101: various single doses, administered to various cohorts
  Interventions: Drug: DDN-A-0101 (SAD)
- Experimental: DDN-A-0101 for PART 2 (Experimental): DDN-A-0101: various multiple doses, administered to various cohorts
  Interventions: Drug: DDN-A-0101 (MAD)
- Placebo Comparator: Placebo for PART 1 (Placebo Comparator): DDN-A-0101 matching placebo: various single doses, administered to various cohorts
  Interventions: Drug: Placebo (SAD)
- Placebo Comparator: Placebo for PART 2 (Placebo Comparator): DDN-A-0101 matching placebo: various multiple doses, administered to various cohorts
  Interventions: Drug: Placebo (MAD)

INTERVENTIONS:
Drug: DDN-A-0101 (SAD) — Investigational drug
  * Development name: DDN-A-0101
  * Main ingredient and content: DDN-A-0101 (Houttuynia cordata dry extract, 150.0 mg)
  * Formulation and properties: Light brown circular film coating tablet
  * Storage method: airtight container, stored at room temperature (1-30 degree celsius)
  * Administration method: single dose oral administration (300, 600, 900, 1200, 1500 mg)
  * Expiration date: 36 months from the date of manufacture
  Arms: Experimental: DDN-A-0101 for PART 1
Drug: DDN-A-0101 (MAD) — Investigational drug
  * Development name: DDN-A-0101
  * Main ingredient and content: DDN-A-0101 (Houttuynia cordata dry extract, 150.0 mg)
  * Formulation and properties: Light brown circular film coating tablet
  * Storage method: airtight container, stored at room temperature (1-30 degree celsius)
  * Administration method: repeated oral administration (150, 300, 450, 600 mg, 2 times/day, 2 weeks of repeated administration)
  * Expiration date: 36 months from the date of manufacture
  Arms: Experimental: DDN-A-0101 for PART 2
Drug: Placebo (SAD) — Placebo drug
  * Development name: placebo of DDN-A-0101
  * Formulation and properties: Light brown circular film coating tablet
  * Storage method: airtight container, stored at room temperature (1-30 degree celsius)
  * Administration method: single dose oral administration (300, 600, 900, 1200, 1500 mg)
  * Expiration date: 36 months from the date of manufacture
  Arms: Placebo Comparator: Placebo for PART 1
Drug: Placebo (MAD) — Placebo drug
  * Development name: placebo of DDN-A-0101
  * Formulation and properties: Light brown circular film coating tablet
  * Storage method: airtight container, stored at room temperature (1-30 degree celsius)
  * Administration method: repeated oral administration (150, 300, 450, 600 mg, 2 times/day, 2 weeks of repeated administration)
  * Expiration date: 36 months from the date of manufacture
  Arms: Placebo Comparator: Placebo for PART 2

SUMMARY:
The study is a Phase I, randomized double-blind, placebo-controlled, single and multiple dosing, dose-escalation study of the oral administration of DDN-A-0101 in healthy adults and elderly subjects

DETAILED DESCRIPTION:
The study includes two Parts; Part1 includes single ascending dose study (SAD) and Part2 includes multiple ascending dose study (MAD). Approximately 50 subjects will be enrolled in the SAD and MAD respectively. New subjects will be recruited for each cohort in both Parts. The SAD Part will include 5 dose levels (S1, S2, S3, S4, S5) and cohort S3 will proceed to food effect cohort. The MAD Part will include 5 dose levels (M1, M2, ME, M3, M4) and cohort ME will be performed in the elderly group.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a healthy adult over 19 years of age and under 65 years of age*.

   *For cohort ME (senior aged person), over 65 years old and under 75 years old a healthy volunteer
2. As a result of the body measurement at the time of screening, the subject has the body weight of 55.0 kg or more and 90.0 kg or less, and the body mass index (BMI) is 18.0 kg/m2 or more and 27.0 kg/m2 or less.
3. The subject who has listened to and listened to sufficient explanations of this clinical trial and voluntarily decided to participate in writing to faithfully implement the compliance with the clinical trial.

Exclusion Criteria:

1. The subject with a history of clinically significant cardiovascular system, respiratory system, kidney, endocrine system, blood system, digestive system, central nervous system, urinary system, musculoskeletal system, psychiatric disease (mood disorders, obsessive-compulsive disorders, etc.) or malignancies (but can be registered if the past history of complete recovery does not affect the current health condition).
2. The subject with a history of gastrointestinal diseases (such as Crohn's disease, ulcers, acute or chronic pancreatitis, hypothyroidism, anaphylaxis, etc.) or gastrointestinal operations (except simple appendectomy or hernia) that may affect the absorption of clinical trials drugs.
3. The subject diagnosed with peptic ulcer, esophageal disease, and Zollinger-Ellison syndrome within 90 days prior to clinical trial drug administration and have been treated or have a medical history or symptoms clinically suspicious of it.
4. The subject showing the following values in the laboratory test results.

   * Blood aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level > 1.5 times normal upper limit
   * Blood Total bilirubin level > 1.5 times normal upper limit
   * Blood creatine phosphokinase (CPK) level > 1.5 times normal upper limit
   * Positive serum epidemiological test results (human immunodeficiency virus (HIV) Ag/Ab, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) Ab, Syphilis regain test)
   * Chronic kidney disease epidemiology collaboration (CKD-EPI) equation calculated creatine cleaning rate: < 60 mL/min/1.73 m2
5. The subject with significant abnormalities in neurological examinations conducted during screening visits.
6. The subject who showed systolic blood pressure ≥ 150 mmHg or < 90 mmHg, diastolic blood pressure ≥ 100 mmHg or < 50 mmHg in blood pressure measured from the upper left after resting for at least 5 minutes at the time of screening.
7. The subject with clinically significant allergic diseases (excluding mild allergic rhinitis that does not require administration)
8. The subject who have a history of drug abuse or are positive for an abuse drug in a urine screening test.
9. The subject who have a history of hypersensitivity reactions to drugs of the same class as the main ingredient and component components of clinical trial drugs.
10. The subject who have received medications from other clinical trials and biological equivalence trials within 6 months of the start of administration of clinical trials.
11. The subject who took metabolic enzyme-induced and inhibitory drugs such as barbital drugs within 30 days prior to administration of clinical trial drugs.
12. The subject who have donated whole blood within 60 days prior to administration of clinical trial drugs or volunteers who have donated or received component blood within 20 days prior to administration of clinical trial drugs.
13. The subject who took over-the-counter drugs or herbal medicines within 14 days of clinical trial administration, or took over-the-counter drugs, health functional foods, or vitamins within 7 days (but may participate in clinical trials if it is deemed that the results of the clinical trial are not affected by the examiner's judgment).
14. The subject who cannot prohibit the administration of the following drugs during the clinical trial period from 8 weeks before the scheduled date of the first administration of the drug for clinical trial.

    * Dementia medications, cognitive enhancers, choline agonists, anti-choline agonists, anti-Parkinson drugs
    * Medicines/supplements/health functional foods and other cosmetics (shampoo, lotion, etc.) containing Houttuynia cordata extract, the main ingredient of this clinical trial drug
    * Medicines or health functional foods with similar indications to other clinical medicines (e.g., extracts derived from ginkgo leaves, etc.)
15. The subject who consumed grapefruit-containing food (one grapefruit or more than 200 ml of grapefruit juice) within 7 days prior to administration of clinical trial drugs.
16. The subject who are forced to consume caffeine (coffee, green tea, etc. >5 cups/day) continuously or consume caffeine-containing food 24 hours before hospitalization during the clinical trial period.
17. The subject who are unable to drink alcohol continuously (alcohol > 210 g/shareholder) or abstain from drinking during clinical trials 24 hours before hospitalization.
18. The subject who cannot smoke excessively (tobacco > 10 skins/day) or quit smoking during the clinical trial period from 24 hours before hospitalization
19. The subject who is pregnant or breast-feeding.
20. The subject who do not agree to use one or more medically acceptable forms of contraception during the pre-clinical period and until at least 90 days after the last clinical trial administration, and those who do not agree to donate sperm or eggs until at least 90 days after the last clinical trial administration. Medically acceptable forms of contraception are as follows.

    * Use of an intrauterine device with proven pregnancy failure rates in the person or partner
    * Use both blocking contraceptives (for male or female use) and spermicide
    * Surgery by yourself or your partner (vasectomy, salpingectomy/ligation, hysterectomy)
21. The subject with a history of suicidal behavior and/or ongoing suicidal ideation following C-SSRS evaluation when screening.
22. The subject deemed unsuitable for participation in clinical trials due to other reasons other than the criteria for exclusion above.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of DDN-A-0101 by monitoring vital signs | through study completion (up to Day 12 for SAD test, Day 25 for MAD test)
  Systolic, diastolic blood pressure (mmHg) measurement to assess vital signs after DDN-A-0101 administration
Assessment of safety and tolerability of DDN-A-0101 by monitoring vital signs | through study completion (up to Day 12 for SAD test, Day 25 for MAD test)
  Pulse rate (bpm) measurement to assess vital signs after DDN-A-0101 administration
Assessment of safety and tolerability of DDN-A-0101 by monitoring vital signs | through study completion (up to Day 12 for SAD test, Day 25 for MAD test)
  Body temperature (°C) measurement to assess vital signs after DDN-A-0101 administration
Assessment of safety and tolerability of DDN-A-0101 by monitoring ECG | through study completion (up to Day 12 for SAD test, Day 25 for MAD test)
  12-ECG electrocardiogram test includes measurement of P-wave (reflecting atrial depolarization), QRS complex (reflecting depolarization of ventricles) and QT interval (reflecting the total duration of ventricular depolarization and repolarization
Assessment of safety and tolerability of DDN-A-0101 by C-SSRS measurement | through study completion (up to Day 12 for SAD test, Day 25 for MAD test)
  Columbia-suicide severity rating scale (C-SSRS) includes the measurement of the incidences and severity of suicidal thoughts
Assessment of safety and tolerability of DDN-A-0101 by laboratory safety tests | through study completion (up to Day 12 for SAD test, Day 25 for MAD test)
  Laboratory safety tests include hematologic test for white blood cell count
Assessment of safety and tolerability of DDN-A-0101 by laboratory safety tests | through study completion (up to Day 12 for SAD test, Day 25 for MAD test)
  Laboratory safety tests include blood chemistry test for measurement of aspartate aminotransferase (AST) and alanine aminotransferase (ALT) (unit/liter)
Assessment of safety and tolerability of DDN-A-0101 by laboratory safety tests | through study completion (up to Day 12 for SAD test, Day 25 for MAD test)
  Laboratory safety tests include urine test for measurement of albumin/creatinine ratio (mg/g)
Assessment of pharmacokinetics of Quercitrin, an indicator of of DDN-A-0101 in plasma | up to 48 hour after intervention
  Area under curve (AUC) in plasma
Assessment of pharmacokinetics of Quercitrin in plasma | up to 48 hour after intervention
  Maximum concentration (Cmax) in plasma
Assessment of pharmacokinetics of Quercitrin in plasma | up to 48 hour after intervention
  Time to peak drug concentration (Tmax) in plasma
Assessment of pharmacokinetics of Quercitrin in plasma | up to 48 hour after intervention
  Half-life in plasma
Assessment of pharmacokinetics of Quercitrin in plasma | up to 48 hour after intervention
  Clearance (CL/F) in plasma
Assessment of pharmacokinetics of Quercitrin in plasma | up to 48 hour after intervention
  Volume of distribution (V/F) in plasma
Assessment of pharmacokinetics of Quercitrin in plasma | up to 48 hour after intervention
  Peak to trough fluctuation ratio (PTF) in plasma
Assessment of pharmacokinetics of Quercitrin in plasma | up to 48 hour after intervention
  Accumulation index (AI) in plasma
Assessment of pharmacokinetics of Quercitrin in urine | up to 48 hour after intervention
  Total amount of Quercitrin excreted in urine (Ae)
Assessment of pharmacokinetics of Quercitrin in urine | up to 48 hour after intervention
  Percentage of Quercitrin excreted in urine (fe)
Assessment of pharmacokinetics of Quercitrin in urine | up to 48 hour after intervention
  Renal clearance (CL) of Quercitrin

SECONDARY OUTCOMES:
Assessment of pharmacodynamics of DDN-A-0101 for PART2 MAD test | up to 24 hour after intervention
  Maximum Effect (Emax) on p-Tau181, C-reactive protein, Interleukin-1 beta, Brain-derived neurotrophic factor
Assessment of pharmacodynamics of DDN-A-0101 for PART2 MAD test | up to 24 hour after intervention
  Area under the effect curve (AUEC) on p-Tau181, C-reactive protein, Interleukin-1 beta, Brain-derived neurotrophic factor

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, Doctor, Principal Investigator — Seoul National University College of Medicine and Hospital
Locations (1):
- Seoul National University College of Medicine and Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No